CLINICAL TRIAL: NCT02008266
Title: Case Study of the Treatment of Early Rheumatoid Arthritis in Algerian Patients in Both the Private and Public Healthcare Sectors.
Brief Title: Study of the Treatment of Algerian Patients With Early Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25384
Record Dates: First submitted 2013-11-27; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis

SUMMARY:
This non-interventional, descriptive, cross-sectional and multicenter study will examine the treatment of rheumatoid arthritis progressing for less than two years in the Algerian population. Current drug therapy as well as disease status and patient function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis progressing for < 2 years.

Exclusion Criteria:

* Rheumatoid arthritis progressing for < 3 months.
* Rheumatoid arthritis onset at < 18 years of age.
* Participation in another clinical study.
* Rheumatoid arthritis related connective tissue disorder.
* Any neuropsychological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis that has been progressing for > 3 months and < 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Describe medications used in the treatment of rheumatoid arthritis with < 2 years' progression. | Single observational visit [Day 1]

SECONDARY OUTCOMES:
Measure disease activity using DAS 28 assessment. | Single observational visit [Day 1]
Assess joint damage using the modified SHARP method. | Single observational visit [Day 1]
Assess functional status of patients using the Health Assessment Questionnaire (HAQ). | Single observational visit [Day 1]

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche